CLINICAL TRIAL: NCT02427477
Title: A Comparison of Two Daily Disposable Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-5698
Record Dates: First submitted 2015-04-22; First posted 2015-04-28 (Estimated); Results first posted 2016-06-13 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2016-07

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- senofilcon A/ delefilcon A/ senofilcon A (Experimental): Subjects were randomized to one two lens wear sequences. Subjects randomized to this sequence first wore the senofilcon A contact lens, then wore the delefilcon A contact lens second and then wore the senofilcon A contact lens third.
  Interventions: Device: senofilcon A; Device: delefilcon A
- delefilcon A/senofilcon A/ delfilcon A (Active Comparator): Subjects were randomized to one two lens wear sequences. Subjects randomized to this sequence first wore the delefilcon A contact lens then wore the senofilcon A contact lens second and then wore the Control lens delefilcon A contact lens third.
  Interventions: Device: senofilcon A; Device: delefilcon A

INTERVENTIONS:
Device: senofilcon A — Subjects will wear the contact lenses in both eyes for seven days
  Other Names: senofilcon A Prototype
Device: delefilcon A — Subjects will wear the contact lenses in both eyes for seven days
  Other Names: Dailies Total 1

SUMMARY:
Approximately 120 subjects will be comparing two soft contact lenses for one week each.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read, understand, and sign the Statement of Informed Consent, and receive a fully executed copy of the form.
2. The subject must be appear able and willing to adhere to instruction set forth in this clinical protocol.
3. The subject be between (and including) 18 and 39 years of age.
4. The subject must be an adapted wearer of spherical soft contact lenses in both eyes. That is, the subject must wear their habitual lenses at least five (5) days per week and eight (8) hours per day worn for at least 30 days immediately preceding the study.
5. The subject's vertex corrected spherical equivalent distance refraction must be in the range of -0.50 to -6.00 D in each eye.
6. The subject must have best corrected visual acuity of 20/25 or better in each eye.

Exclusion Criteria:

1. Currently pregnant or breastfeeding (subjects who become pregnant during the study will be discontinued).
2. Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
3. Any autoimmune disease or use of any medication, which may interfere with contact lens wear.
4. Entropoin, Ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, or aphakia.
5. Any previous, or planned ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, etc.)
6. Any grade 3 or greater slit lamp findings (e.g. edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related inflammatory event (e.g. past peripheral ulcer or round scar), or any other ocular abnormality that may contraindicate contact lens wear.
7. Any ocular infection.
8. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
9. Monovision, multifocal, toric, or extended wear contact lens correction.
10. Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
11. History of binocular vision abnormality or strabismus.
12. Any infectious disease (e.g. hepatitis, tuberculosis) or contagious immunosuppressive disease (e.g. HIV) by self-report.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Montgomery, Alabama
  - Jacksonville Beach, Florida
  - Longwood, Florida
  - Winter Park, Florida
  - Westerville, Ohio
  - Salem, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 120 subjects were enrolled into this study. All enrolled subjects were dispensed a study lens. Of the dispensed subjects 1 was discontinued from the study and 119 subjects completed the study.
Groups:
- Senofilcon A / Delefilcon A/ Senofilcon A: Subjects were randomly assigned to one of two lens sequences, over three lens wear periods. Subjects randomized to this sequence first wore the senofilcon A contact lens, then wore the delefilcon A contact lens second and then wore the senofilcon A contact lens third.
- Delefilcon A / Senofilcon A / Delefilcon A: Subjects were randomly assigned to one of two lens sequences, over three lens wear periods. Subjects randomized to this sequence first wore delefilcon A contact lens, then wore the senofilcon A second and then wore the delefilcon A contact lens third.
Period: Period 1
Arm/Group | Senofilcon A / Delefilcon A/ Senofilcon A | Delefilcon A / Senofilcon A / Delefilcon A
Started | 60 | 60
Completed | 59 | 60
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Period 2
Arm/Group | Senofilcon A / Delefilcon A/ Senofilcon A | Delefilcon A / Senofilcon A / Delefilcon A
Started | 59 | 60
Completed | 59 | 60
Not Completed | 0 | 0
Period: Period 3
Arm/Group | Senofilcon A / Delefilcon A/ Senofilcon A | Delefilcon A / Senofilcon A / Delefilcon A
Started | 59 | 60
Completed | 59 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that randomized to one of two sequences of lens wear.
Groups:
- Senofilcon A / Delefilcon A / Senofilcon A; Delefilcon A / Senofilcon A / Delefilcon A: All subjects that randomized to receive this sequence and were dispensed a study lens.
- Total: Total of all reporting groups
Arm/Group | Senofilcon A / Delefilcon A / Senofilcon A | Delefilcon A / Senofilcon A / Delefilcon A | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.6 (6.14) | 27.6 (4.97) | 28.0 (5.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 38 | 80
  Male | 18 | 22 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 3 | 14
  White | 47 | 52 | 99
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Subjective Overall Comfort
Description: Subjective Overall Comfort was evaluated using the Contact Lens User Experience Comfort scores (CLUE). CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response.
Time Frame: 1-week Follow-up
Population: The Analysis population includes subjects that completed all study visits without a major protocol deviation. Due to the study design the number of observations analyzed is larger than the number of participants. This is due to the fact that some subjects wore senofilcon A twice while some subjects wore delefilcon A twice (see Participant Flow).
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Observations
Groups:
- Senofilcon A: Subjects that received the senofilcon A contact lens in at least one of the three study periods.
- Delefilcon A: Subjects that received the delefilcon A contact lens in at least one of the three study periods.
Arm/Group | Senofilcon A | Delefilcon A
Number analyzed (Participants) | 119 | 119
Number analyzed (Observations) | 178 | 179
units on a scale | 75.5 (28.12) | 70.8 (28.60)

2. Primary Outcome: Subjective Overall Vision
Description: Subjective Overall Vision was evaluated using the Contact Lens User Experience Vison scores (CLUE). CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response.
Time Frame: 1-week Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Observations
Arm/Group | Senofilcon A | Delefilcon A
Number analyzed (Participants) | 119 | 119
Number analyzed (Observations) | 178 | 179
units on a scale | 75.3 (22.04) | 72.1 (24.05)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study- approximately 1 month.
Arm/Group | Senofilcon A | Delefilcon A
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/120
Other Adverse Events (participants affected / at risk) | 0/120 | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less